CLINICAL TRIAL: NCT06120790
Title: Investigation of a 3 oz Water Protocol on Patients With Tracheostomies
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Miguel Escalon, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-23-00005
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Tracheostomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Tracheostomies: Patients with openings in their airways (i.e. tracheostomies)
  Interventions: Other: 3 Oz water screen

INTERVENTIONS:
Other: 3 Oz water screen — Patient will consume 3 oz of water continuously without stopping and then will be monitored for one minute post completion. Patient will complete this twice in the same session.

SUMMARY:
Examining the validity of a novel 3 oz protocol in patients with tracheostomies as compared to the gold standard of instrumental swallow assessments (Flexible Endoscopic Evaluation of the Swallow or Modified Barium Swallow Study).

DETAILED DESCRIPTION:
The purpose of this research study is to determine if a 3 oz water screening protocol is an effective screen for patients with openings in their airways (i.e. tracheostomies). This procedure is already in use for many different populations and is particularly useful for clinicians who want to understand who is at risk for having food or liquid enter the lungs while eating or drinking (i.e. aspiration).

ELIGIBILITY:
Inclusion Criteria:

* Has a tracheostomy
* Able to remain alert for testing
* Not on a modified diet for pre-existing dysphagia
* No head of bed restrictions
* Not NPO by physician for any reason other than possible dysphagia
* At least 18 years old

Exclusion Criteria:

* Does not have a tracheostomy
* Unable to remain alert for testing
* On a modified diet due to pre-existing dysphagia
* Head of bed restrictions for greater than or equal to 30 degrees
* NPO by physician for reasons other than possible dysphagia
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a tracheostomy (dysphagia).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Swallow screen | End of participation study within 7 days of enrollment
  Swallow screen measured as pass/fail for presence or absence of aspiration
Penetration Aspiration Scale Score | End of participation study within 7 days of enrollment
  The penetration aspiration scale (PAS) is a validated measure used by trained blinded clinicians to assign ratings of safety to swallowing bolus trials. The PAS is an 8-point, equal-appearing interval scale (8 being best; 1 being worst) to describe penetration and aspiration events. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled. Higher scores indicate better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Escalon, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Proposals should be directed to miguel.escalon@mountsinai.org.